CLINICAL TRIAL: NCT06492915
Title: A Phase Ⅱ Study of Chiauranib Plus Albumin-paclitaxel and Gemcitabine as First-line Therapy in Patients With Locally Advanced or Metastatic Pancreatic Ductal Adenocarcinoma
Brief Title: Chiauranib in Patients With Locally Advanced or Metastatic Pancreatic Ductal Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chipscreen Biosciences, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAR205
Record Dates: First submitted 2024-06-27; First posted 2024-07-09 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-07

CONDITIONS: Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — chiauranib; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Chiauranib plus albumin-paclitaxel and gemcitabine (Experimental): Participants received Chiauranib oral administration once daily. Albumin-paclitaxel Injection and Gemcitabine Injection administered intravenously on Days 1, 8 and 15 of each 28-day cycle.
  Interventions: Drug: Chiauranib; Drug: Albumin-paclitaxel Injection; Drug: Gemcitabine Injection

INTERVENTIONS:
Drug: Chiauranib — Chiauranib, 25 mg, 35 mg or 50 mg, oral administration once daily
Drug: Albumin-paclitaxel Injection — Albumin-paclitaxel Injection, 125 mg/m^2 administered intravenously on Days 1, 8 and 15 of each 28-day cycle
Drug: Gemcitabine Injection — Gemcitabine Injection, 1000 mg/m^2 administered intravenously on Days 1, 8 and 15 of each 28-day cycle

SUMMARY:
Chiauranib , which simultaneously targets against VEGFR/Aurora B/CSF-1R, several key kinases involved in tumor angiogenesis, tumor cell mitosis, and chronic inflammatory microenvironment.

DETAILED DESCRIPTION:
Chiauranib is a novel orally active multi-target inhibitor that simultaneously inhibits the angiogenesis-related kinases (VEGFR2, VEGFR1, VEGFR3, PDGFRa and c-Kit), mitosis-related kinase Aurora B and chronic inflammationrelated kinase CSF-1R in a high potency manner with the IC50 at a single-digit nanomolar range. In particular, Chiauranib showed very high selectivity in the kinase inhibition profile with little activity on off-target non-receptor kinases, proteins, GPCR and ion channels, indicative of a better drug safety profile in terms of clinical relevance.

This study is a phase II, single arm, open label, multi-center study to evaluate the efficacy and safety of chiauranib plus albumin-paclitaxel and gemcitabine as first-line therapy in patients with locally advanced or metastatic pancreatic ductal adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign the written informed consent form.
2. Age 18-75 years on the day of signing the informed consent form, male or female.
3. Histologically or cytologically confirmed unresectable locally advanced or metastatic pancreatic ductal adenocarcinoma.
4. No prior systemic therapy for unresectable locally advanced or metastatic pancreatic ductal adenocarcinoma. Subjects who have received prior induction chemotherapy, concurrent radiotherapy, or adjuvant/neoadjuvant chemotherapy with curative intent, the interval of recurrence or metastasis must be at least 6 months after the last treatment.
5. At least one measurable lesion according to RECIST v1.1. Previously irradiated lesions should not be selected as target lesions unless the previously irradiated lesion as the only measurable lesion and is unequivocally progressive based on imaging.
6. ECOG score 0 or 1.
7. Life expectancy≥3 months.
8. Major organ functions meet the following criteria: Hematology: hemoglobin≥90g/L, absolute neutrophil count (ANC) ≥1.5×10^9/L, platelets≥100×10^9/L(no haematopoietic growth factors or blood transfusions and other medications considered by the investigator to be corrective therapy, within 2 weeks before enrollment). Biochemistry: serum creatinine≤1.5×ULN, total bilirubin≤1.5×ULN, AST/ALT≤2.5×ULN (≤5×ULN for patients with hepatic metastasis). Coagulation Function: INR < 1.5×ULN.

Exclusion Criteria:

1. Histological or cytological confirmed other pathological types, such as acinar cell carcinoma, neuroendocrine carcinoma, pancreablastoma, etc.
2. Previous received Aurora kinase inhibitors or systemic treatment of VEGF/VEGFR inhibitors such as bevacizumab, sorafenib, sunitinib, amlotinib, apatinib, and endostar.
3. Previous radiation therapy, chemotherapy, immunotherapy, targeted therapy within 28 days prior to the first dose. Traditional Chinese medicine (except for Chinese herbal medicine) witn anti-malignancy effect judged by the investigator within 14 days prior to the first dose.
4. Presence of active or untreated brain metastases, meningeal metastases, spinal cord compression, or molluscum contagiosum disease during the screening period. However, enrolment is permitted for subjects who meet the following requirements and have measurable lesion outside the CNS: asymptomatic after treatment and stable on imaging for at least 4 weeks prior to the first dose (e.g., no new or enlarging brain metastases) and have been off systemic glucocorticosteroids and anticonvulsant medications for at least 2 weeks prior to the first dose.
5. Presence of clinically symptomatic pleural effusion, pericardial effusion or ascites requiring frequent drainage (≥1 time/month) during the screening period.
6. Major surgery (craniotomy, thoracotomy, or laparotomy) or serious unhealed wounds, ulcers, or fractures within 4 weeks prior to the first dose. Needle biopsy or other minor surgery (except for intravenous infusion) within 7 days prior to the first dose.
7. Significant arterial/venous thrombotic events within 6 months prior to first dose, such as deep vein thrombosis and pulmonary embolism. Superficial vein thrombosis without safety risk judged by the investigator is permitted.
8. Cardiac dysfunction or clinically meaningful cardiovascular disease, including: (1)New York Heart Association (NYHA) grade II or higher congestive cardiac failure, unstable angina pectoris, and/or myocardial infarction within the 6 months prior to the first dose of the investigational drug, clinically significant arrhythmia unable to be controlled with medical treatment or left ventricular ejection fraction (LVEF) < 50% at screening. (2)Primary cardiomyopathies (e.g., dilated cardiomyopathy, hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, restrictive cardiomyopathy, indeterminate cardiomyopathy). (3)Clinically significant history of prolonged QTc interval, or QTcF interval >470ms for females or >450 ms for males during the screening period. (4)Coronary heart disease with symptoms requiring medication. (5)Documentation of hypertension treatment with≥3 antihypertensive medications simultaneously within 14 days before the first dose of medication or systolic blood pressure≥140 mmHg and/or diastolic blood pressure≥90 mmHg during the screening period (resting state, measured approximately every 5 minutes, averaged after three consecutive measurements, rounded to the nearest integer). (6)History of hypertensive crisis or hypertensive encephalopathy. (7)Other cardiovascular disease judged by the investigator to be unsuitable for enrolment.
9. Active bleeding within 2 months prior to the first dose, or taking anticoagulants, such as warfarin, phenprocoumon (prophylactic low-dose aspirin and low-molecular heparin are permitted) during the screening period, or at high risk of bleeding judged by the investigator during screening period (e.g., esophageal varix associated with bleeding risk, locally active ulcer lesions, positive fecal occult blood that can not exclude gastrointestinal bleeding, intermittent haemoptysis) .
10. Presence of significant gastrointestinal abnormalities during the screening period that may interfere with drug intake, transit or absorption (e.g. inability to swallow, chronic diarrhoea, post-small bowel resection or total gastrectomy), according to the investigator's judgment.
11. History of gastrointestinal perforation and/or fistula, peptic ulcer disease, intestinal obstruction (including incomplete intestinal obstruction that requires parenteral nutrition), or biliary obstruction within 6 months prior to the first dose.
12. History of other malignant tumors within 3 years prior to the first dose, except for those treated with expected curative outcomes, such as basal cell carcinoma, squamous cell carcinoma of the skin, superficial bladder cancer, carcinoma in situ of the cervix, ductal carcinoma in situ of the breast, localized prostate cancer, and papillary thyroid microcarcinoma.
13. For urine protein≥2+ by urinalysis during the screening period, a 24-hour urine protein quantification test should be performed. The subject cannot be enrolled if the quantified urine protein is≥1g/24 h. If the quantified urine protein is <1 g/24 h, the subject can still be enrolled.
14. Presence of peripheral neuropathy of CTCAE v5.0 criteria, Grade 2 or higher.
15. Known contraindications to albumin-paclitaxel and gemcitabine chemotherapy (see descriptions for albumin-paclitaxel and gemcitabine).
16. Adverse effects of prior antineoplastic therapy that have not returned to ≤grade 1 of CTCAE v5.0 criteria (except for alopecia without safety risk judged by the investigator and laboratory tests specified in Inclusion Criterion 8).
17. Presence of clinically active haemoptysis, active diverticulitis during the screening period.
18. Presence of active tuberculosis during the screening period. Suspected subjects should be excluded by a combination of chest imaging, sputum, and through clinical signs and symptoms.
19. Presence of active hepatitis of positive HBsAg with positive viral replication or positive HBcAb with positive viral replication during the screening period. Positive HCV-Ab with positive viral replication. Positive of HIV. Active syphilis infection (syphilis-specific antibody and nonspecific antibody positive). (Note: Priority for qualitative detection and quantitative detection of viral replication when needed).
20. Previous or screening chest imaging showing the presence of interstitial lung disease or pulmonary fibrosis or non-infectious pneumonitis requiring treatment, and immune-associated pneumonia after previous treatment with PD-1/PD-L1 inhibitor.
21. Active infection during the screening period, including systemic anti-infective therapy requiring oral or intravenous infusion within 2 weeks prior to the first dose, unexplained fever (≥38°C, except for tumor causes judged by the investigator) during the screening period.
22. Screening period or history of allogeneic organ transplantation and allogeneic haematopoietic stem cell transplantation.
23. Unexplained weight loss of 5% or more between signing the ICF and the first dose.
24. NRS pain score 4 after analgesic medication during the screening period.
25. Severe central nervous system or psychiatric illness during the screening period.
26. Pregnant or lactating females. Female subjects of childbearing potential or male subjects whose partners of childbearing potential are unable or unwilling to use effective contraception (e.g., IUDs, Subcutaneous implant, sterilisation, long-acting contraceptive injections, compound of short-acting oral contraceptives, etc.) from 7 days prior to the first dose until 6 months after the end of treatment. Female subjects of childbearing potential must have a blood pregnancy test negative witnin 7days prior to the first dose.
27. During the screening period, the investigator deems other conditions unsuitable for participation in this trial, such as clinically unacceptable worsening symptoms or signs of pancreatic cancer progression, comorbidities, concurrent treatments, or any laboratory abnormalities that may interfere with the assessment of efficacy and safety outcomes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
PFS | From the first dose to disease progression or end of study, an average of 1 year
  Progression free survival

SECONDARY OUTCOMES:
ORR | From the first dose to disease progression or end of study, an average of 1 year
  Objective Response Rate
DCR | From the first dose to disease progression or end of study, an average of 1 year
  Disease control rate
DoR | From the first dose to disease progression or end of study, an average of 1 year
  Duration of Response
TTR | From the first dose to disease progression or end of study, an average of 1 year
  Time to Response
OS | From the first dose to death or end of study, an average of 1.5 years
  Overall survival
Adverse events | From the enrollment until 28 days after the last dose
  Incidence of adverse events (defined by the Common Terminology Criteria for Adverse Events version 5.0 (CTCAEV5.0))
Time to maximum concentration (Tmax) | Days 15, 28 during Cycle 1, thereafter once every 8 weeks subsequent cycles, an average of 1 year
  PK Profile
Maximum plasma concentration (Cmax) | Days 15, 28 during Cycle 1, thereafter once every 8 weeks subsequent cycles, an average of 1 year
  PK Profile
Area under the plasma concentration-time curve (AUC0-t) | Days 15, 28 during Cycle 1, thereafter once every 8 weeks subsequent cycles, an average of 1 year
  PK Profile

CONTACTS AND LOCATIONS:
Overall Officials: Xianjun Yu, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No